CLINICAL TRIAL: NCT04126837
Title: Accelerated Nursing Branch for the Diagnosis and Treatment of Ankle and Foot Injuries in Emergency Department: Preliminary Pilot Study
Brief Title: Ankle Trauma: an Emergency Nurse Assessment Study
Acronym: ATENA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 38RC19.200
Record Dates: First submitted 2019-10-01; First posted 2019-10-15 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Ankle Injuries; Foot Injuries; Diagnosis; Treatment
Keywords: Ankle; Foot; Injuries; Ottawa Rules; nurse
MeSH Terms: conditions — Ankle Injuries; Foot Injuries; Disease; Wounds and Injuries | interventions — Therapeutics; Emergency Service, Hospital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient admitted for Ankle and foot injuries (Other): Diagnosis and treatment of Ankle and foot injuries by an accelerated nursing branch in emergency department
  Interventions: Other: Diagnosis and treatment

INTERVENTIONS:
Other: Diagnosis and treatment — Monocentric, Prospective and Biomedical Research excluding Health Product
  Other Names: Assessment of an accelerated nursing branch for the diagnosis and treatment of ankle and/or foot injuries in emergency department.

SUMMARY:
The ankle and/or foot injuries incidence is high. Lateral ankle sprains are most common diagnosis, while fractures represent less than 15% of final diagnosis. Ankle and/or foot injuries are associated with significant morbidity in terms of pain and chronic instability. The societal cost of these injuries is significant mainly related to hospital care and sick-leave. In summary ankle and/or foot injuries are very frequent reason for emergency admission.

The study hypothesis is that an accelerated nursing care system for traumatized ankle and/or foot patients is feasible and allows patients to be cared for in accordance to current medical recommendations. Such a branch should be followed by a return to work and sports within a time frame consistent with the literature. The duration of patient management in emergency department should be short, less than that observed in a historical cohort. Finally patient satisfaction should be high. In the medium term, the implementation of an accelerated nursing branch for the diagnosis and treatment of ankle and/or foot injuries should contribute to effective care and reduction of over activity in emergency departments.

DETAILED DESCRIPTION:
The incidence of ankle and/or foot injuries is high. Lateral ankle sprains are the most common diagnosis, while fractures represent less than 15% of the final diagnosis. Ankle and/or foot injuries are associated with significant morbidity in terms of pain and chronic instability. The societal cost of these injuries is significant mainly related to hospital care and sick-leave. Ankle and/or foot injuries are very frequent reason for emergency admission.

The aim of this study is to assess the accelerated nursing branch for the diagnosis and treatment of ankle and/or foot injuries in emergency department.

Target Follow-Up duration: 1 month (30 days).

The study will be conducted in 3 phases:

1. Training volunteer emergency department nurses. The training course of 10-hours session (2 hours e-learning and 8 hours attendance) will cover all aspects of management of ankle and/or foot injuries (from diagnosis to treatment). The nurses will have at least one year of clinical experience in emergency department. This training will be conducted by medical experts (emergency doctor, radiologist and orthopedist ). At the end of the training a formative assessment both theoretical and practical will be carried out with participants.

   The following intervention will be performed by emergency nurses:
   * Pain intensity assessment
   * Record of the trauma mechanism and history of the patient
   * Ottawa rules and clinical examination
   * Radiographic prescription and interpretation
   * Prescription and interpretation of additional examination
   * Foot and Ankle Survey (FAO)
   * Evaluation of ankle joint function
   * Treatment: medicine prescription, immobilization, physiotherapy…. Following the management of ankle and/or foot injuries patients by a nurse, every working day a systemic review of the emergency file including X-rays performed will be carried out by a medical staff composed of an emergency doctor, an orthopedist and a radiologist. This review will be done every morning in the emergency department.
2. Enroll patients admitted to the emergency department for ankle and/or foot injuries. The ability of trained nurses to treat these traumas will be assessed.
3. Phone follow-up of patient after one month to collect data: the date of return to work or sports, patient satisfaction and possible consultation (by a physician, an orthopedist and/or care consummation).

Two groups of data will be collected: clinical and paraclinical parameters. Clinical parameters: respiratory rate, saturation, blood pressure, heart rate, Glasgow score , weight, size, Numerical Scale ranges of pain , Ottawa rule, treatment, radiography..

Paraclinical parameters: radiography examination, X-ray interpretation, Foot and Ankle Survey(FAS), Evaluation of ankle joint function, patient satisfaction survey, follow-up at one month (30 days).

Outcome measure

The overall adequacy of care will be assessed at the end of the study by a committee of experts whose judgment will be based on the latest medical recommendations. This expert committee will consist of an orthopedic physician, a radiologist, an emergency physician and a quality health executive (nurse) and will make decisions by consensus. These members will be independent of the investigators of the study. The delivered care will be considered globally adequate if it respects the recognized indications of:

* Realization and interpretation of radiography (Ottawa criteria and early radiography service protocol)
* analgesic treatments according to the recommendations of the scientific societies (acetaminophen for EN> 0 +/- WHO step 2 treatment for pain of moderate intensity and WHO step 3 for pain of severe intensity)
* Immobilization: according to the recommendations of the scientific societies: protocol RICE (Rest, Ice,Compression and elevation) immobilization plastered in case of fracture etc.
* Specialist advice: orthopedic opinion if a fracture or other severe pathology is detected

Study design

• Estimation enrollment: 66 participants A sample of 60 patients can be used to estimate an adequate percentage of care tending towards 100% (optimal management defined by the experts), with an accuracy of 5% corresponding to the lower limit of the one-sided confidence interval. 95% (PASS vs 15.0.5., NCSS, LLC, Kaysville, Utah, USA). This is equivalent to establishing 95% non-inferiority using an exact one-sided test with a power of 80% (Normal approximation). A rate of patients lost to follow-up estimated at 10% implies that 66 patients will have to be included.

Analysis:

The main objective of this pilot study is to assess the feasibility of managing ankle or foot trauma by an emergency nurse protocol, describing the percentage of patients who are adequately cared for by this protocol. Statistical methods will therefore be essentially descriptive.

The descriptive analysis will cover all the variables collected. The quantitative parameters for which normality has been accepted will be described by mean and standard deviation. They will be expressed as median, 25th and 75th percentiles when normality has been rejected. The qualitative parameters will be expressed in numbers and percentages framed by their 95% confidence interval.

Serious Adverse events The individual risk is related to a possible misdiagnosis of the nurse who took care of the patient, requiring a further consultation with a general practitioner or emergency. A systematic re-reading of x-rays by the daily medical staff is planned in working days. Patients will be contacted directly by an emergency doctor to advise them to consult their treating or specialist doctor, in case of anomaly detected during the re-reading of the radiography and / or a marked adequacy on the immobilization techniques.

In addition, the following adverse events are likely to occur, related to the management of on-trial trauma care:

* Complications related to limb immobilization (venous thrombosis, eschar, nerve and/or vascular compression)
* Complications related to analgesics Given the purpose of the research and the low risk associated with the investigation procedures, no monitoring committee and no interim analysis are planned. In the event of a security alert, the expert committee will inform the promoter.

In the event of an adverse event considered to be severe by the investigator and possibly involving the health of the subjects, the investigator may stop the study in agreement with the promoter.

ELIGIBILITY:
Inclusion Criteria:

* Isolated Ankle and/or foot Trauma out of dermabrasion
* Admission to emergency department < 48 hours after the trauma
* Written informed consent must be obtained
* For women of childbearing age: effective contraception in place for at least 3 months

Exclusion Criteria:

* X-ray performed before patient admission
* Obvious open fracture
* Ankle fracture or obvious deformation
* Suspicion of polytrauma
* Anterior surgery of the ankle and/or foot
* Excessive alcoholization or intoxication by other psychoactive substances
* Persons unable to communicate in french, with impaired comprehension skills and consciousness (problem with mental health)
* Adults legally protected (under judicial protection, guardianship, or supervision), persons deprived of liberty
* Non-affiliated to the french social security system (or equivalent)
* Pregnant or nursing women
* Patient participating in any interventional clinical reserach study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who have received a diagnosis and treatment in accordance with medical recommendations. | 30 days
  Percentage of patients who have received a diagnosis and treatment by nurse in accordance with medical recommandation

SECONDARY OUTCOMES:
Percentage of patients with diagnosis in accordance with Ottawa rules | 1 day
  Percentage of patients managed by nurse with diagnosis in accordance with Ottawa rules
Description of pain intensity | 1 day
  Pain intensity assessed by a Numerical Scale ranges (0-10) during admission, on arrival in care areas and during discharge
Deadline for return to work and /or sports | 30 days
  delay (number of days) between the trauma and return to work and/ sports
Consummation of care (excluding medicines) | 30 days
  number of possible consultation after emergency discharge and 30 days
Evaluate the time required to manage patients | 30 days
  Mean length of stay (MLD) in emergency department compared to the MLD of a historical cohort of patients admitted to emergency department for ankle and foot injuries
Percentage of refusal in participation of the study | 30 days
  Percentage of patients screened but who refused to participate in the study
Patient satisfaction assessed during discharge and in one month | 1 and 30 days
  Patient satisfaction assessed during discharge and in one month evaluated by visual analog scale (VAS) during discharge and in one month. The VAS scale ranges are: (Not at all satisfied patientwould no longer accept a nurse's care - Completely satisfied patient would accept to be cared for again by a nurse)

CONTACTS AND LOCATIONS:
Overall Officials: Damien VIGLINO, MD,PhD, Principal Investigator — Emergency Department of University Hospital Grenoble; Nicolas TERMOZ MASSON, Bachelor, Study Director — Emergency Department of University Hospital Grenoble; Alexandra BICHET, Bachelor, Study Director — Emergency Department of University Hospital Grenoble
Locations (1):
- Grenoble Alpes University Hospital, Grenoble, Isere, France

IPD SHARING:
Plan to Share IPD: Yes
The international writing and publication rules (The Uniform Requirements for Manuscripts of the ICMJE, April 2010) will be followed. The minimum anonymized source data for performing the statistical analysis will be made public at the time of publication, with the article, or deposited in an appropriate public database. Other anonymized data may be available from the principal investigator upon reasonable request and with the consent of the sponsor.
  In accordance with the French law n ° 2002-303 of March 4th, 2002, the subjects can be informed, at their request, of the overall results of the research. In this study, the investigators commit to individually communicating the overall results to each subject participating in the research by a short (popularized) summary and associated with a copy of the scientific article.
Supporting Information: Study Protocol, SAP
Time Frame: at the time of publication
Access Criteria: The international writing and publication rules (The Uniform Requirements for Manuscripts of the ICMJE, April 2010) will be followed. And In accordance with the French law n ° 2002-303 of March 4th, 2002